CLINICAL TRIAL: NCT00855257
Title: Assessment of Endothelial Vasomotricity After Treatment by Nicotinic Acid in Patients Presenting a Recent Acute Coronary Syndrome.
Brief Title: Assessment of Endothelial Vasomotricity After Treatment by Nicotinic Acid in Acute Coronary Syndrome
Acronym: EVANACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Pr Meyer Elbaz, Rangueil Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-07
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Acid nicotinique; FLOW MEDIATED DILATATION (FMD); HDL-C< 0.4 G/L
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): treatment by acid nicotinique
  Interventions: Drug: Acid Nicotinique
- 2 (Placebo Comparator): Treatment by placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acid Nicotinique
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The investigators' work proposes to evaluate the effectiveness of the Acid Nicotinique (Niaspan®), only molecule currently marketed, ready to raise the plasmatic levels of HDL-c. This effectiveness will be tested among patients having presented recently an acute coronary syndrome. The effectiveness of the molecule will be appreciated versus placebo after randomization.

The technique of evaluation of this effectiveness will be the analysis of the vasodilatation endothelial-dependent measured on the level huméral (by echography high resolution).

The awaited result is an improvement of 2% in value absolute of this vasodilatation between the initial test and the end of study for the patients receiving the acid nicotinic versus those receiving the placebo (3 months of treatment after inclusion). The calculation of the sample necessary to achieve this goal envisages 70 patients led at the end of the study, divided into two groups of treatment (acid nicotinic or Placebo).

Such a result if it were obtained would be higher than that found in studies evaluating the effect on the vasomotricity endothelial statins or inhibitors of the enzyme of conversion.

DETAILED DESCRIPTION:
The pharmacological assumption of responsibility of the coronary disease has rested partially for a few years on the regulation of the inhibitors of the HMG CoA reductase (statins). These drugs initially address to the quantitative anomalies Lipoproteins of low density (LDL cholesterol). The objectives laid down by the national recommendations (obtaining a plasmatic rate < 1gr/l in coronary secondary prevention or among patients at the high vascular risk) or international, implies their broad regulation with the waning of the coronary syndromes. It can exist in addition among many patients of the qualitative or quantitative anomalies of the Lipoproteins of High density (HDL-c) whose correlation to the coronary risk was beforehand largely shown. The anomalies of HDL-c are not very sensitive to the hygieno-dietetic rules.

To intervene on the plasmatic levels of the lipoproteins is thus essential with the improvement of the forecast of the proven coronary patients.

The investigators know since the beginning of the years 1980 (work of Furchgott and Moncada) that the endothelium is a powerful integrator of the vascular risk, in particular in its aspect of regulation vasomotrice.

Methods of investigation of the endothelium were developed on the coronary floor or the level of the peripheral arteries to analyze the vasomotricity endothelial dependent. Among these methods the study of the vasomotricity on the level huméral is validated, largely used and correlated in many tests with the forecast of the patients presenting a high vascular risk.

ELIGIBILITY:
Inclusion Criteria:

* informed consent written of the patient
* Acute coronary syndrome going back to less than 7 days by the rise higher than 0.10 in troponin associated at least one in the following elements:(symptoms of myocardiac ischaemia, appearance of pathological waves Q, disturb repolarisation in connection with an ischaemia (known or under shift of the segment ST).
* HDL - C lower than 0.4 g/l
* FMD < 7%

Exclusion Criteria:

* Antecedents of myopathy induced by a statin or severe reaction of over-sensitiveness to an inhibitor of the HMG CoA réductase (statins).
* Antecedent of family hypercholesterolemia of homozygote type.
* Women pregnant, nursing, likely to be pregnant and not using chemical or mechanical contraception or presenting a positive test of pregnancy blood (b-HCG).
* Subjects whose substitute hormonal treatment or oral contraception was initiated in the 3 previous months Visit 0.
* Active hepatic pathology or hepatocellular insufficiency (doubly of the gammas WP; TGP > 3 times the normal)
* Renal insufficiency engraves with clearance of creatinin < 30 ml/min.
* LDL<0.70gr/l, triglycerides ³ 400 Mg dL (4.52 mmol/L), hbA1c > 8.5%, HDL cholesterol > 0 40g/l.
* Evolutionary cancer
* Use of the following concomitant treatments: insulin, nitrated derivatives
* Antecedents of alcoholism and/or catch dopes during the last year.
* CPK ³ 3 times higher limit of the normal and fraction MB of CPK < 2 times limit higher of the normal than visit 1. If the CK-MB are not available, one will take into account a value of CPK > 3 times the limit higher of the normal and cardiac Troponin (I or T) < 0.10 g/l than visit 1.
* Clinical history of permanent systolic hypotension (NOT < 90 mmHg) or permanent not controlled hypertension (NOT > 200 mmHg gold PAD > 110 mmHg).
* Coronary bridging in the 3 months before inclusion (V1).
* Occurred of fibrillation ventricular, tachycardia ventricular constant (other which RIVETTED), complete and permanent auriculo-ventricular Bloc, which has occurred of auricular fibrillation with a ventricular rate/rhythm not controlled (> 130 bpm), or ventricular rate/rhythm in the 4 weeks preceding visit 1.
* Cerebral vascular accident, severe infection, péricardite acute or any other obviousness of known systemic embolism not controlled
* Hypothyroïdie defined by a rate of TSH > 1,5 times higher limit of the normal
* Serious or unstable conditions psychological or medical which according to the opinion of the investigator, would compromise the safety of the patient or his participation in the study.
* Participation in another clinical trial (other than registers not raising of a biomedical law of research) with treatment the study or having received a treatment the study in the 4 weeks preceding inclusion in the study.
* Patients under supervision or trusteeship or without Social Security cover or impossibility of following the specific procedures of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Measure of endothelial function by high resolution echography in response to nitric agent | Within the first 7 days of ACS and 3 months by treatment with nicotinic acid

SECONDARY OUTCOMES:
Measure of plasmatic CRP, cytokines, lipid level | Within the first 7 days of ACS and 3 months by treatment with nicotinic acid

CONTACTS AND LOCATIONS:
Overall Officials: meyer elbaz, md phd, Principal Investigator — hopital de rangueil service of cardiology
Locations (1):
- Hôpital de Rangueil, Toulouse, France